CLINICAL TRIAL: NCT01231191
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Relationship Between Intraoperative Intravenous Acetaminophen and Postoperative Opioid Avoidance for Ambulatory Surgical Procedures
Acronym: Cadence
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study not funded
Sponsor: University of California, San Diego (Other)
Collaborators: Cadence Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Associate Professor, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IV Acetaminophen
Record Dates: First submitted 2010-10-27; First posted 2010-11-01 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Postoperative Pain; Intraoperative and Postoperative Opioid Requirements
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Acetaminophen (Active Comparator): Intraoperative IV acetaminophen administered
  Interventions: Drug: Intravenous acetaminophen
- IV Placebo (Placebo Comparator): Intraoperative IV normal saline administered
  Interventions: Drug: Intravenous placebo

INTERVENTIONS:
Drug: Intravenous acetaminophen — Acetaminophen 1000 mg administered over 15 minutes intravenously as soon as feasible intraoperatively.
  Arms: IV Acetaminophen
Drug: Intravenous placebo — Normal saline administered over 15 minutes intravenously as soon as feasible intraoperatively.
  Arms: IV Placebo

SUMMARY:
This is a research study to determine if giving acetaminophen intravenously in hte operating room will decrease the number of patients who require additional pain medicine, such as morphine, after surgery in the recovery room.

DETAILED DESCRIPTION:
Primary Specific Aim: To determine if adding an intraoperative dose of intravenous acetaminphen to usual and customary analgesics during ambulatory surgery impacts the proportion of patients remaining opioid-free in the post-anesthesia recovery room.

Hypothesis: Adding an intraoperative dose of intravenous acetaminophen to usual and customary analgesics during ambulatory surgery increases the proportion of patients remaining opioid-free in the post-anesthesia recovery room.

Secondary Specific Aim: To determine if adding an intraoperative dose of intravenous acetaminophen to usual and customary analgesics during amublatory surgery impacts the required doses of additional perioperative analgesics.

Hypothesis: Adding an intraoperative dose of intravenous acetaminophen to usual and customary analgesics during ambulatory surgery decreases the required doses of additional analgesics in both the operating room and post-anesthesia recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing ambulatory surgery under general anesthesia
* Expected postoperative pain to be mild-moderate
* Age 18 years or older
* Have an ASA physical status or 1, 2, or 3

Exclusion Criteria:

* Anticipated peripheral or neuraxial nerve block
* Any physical, mental or medical conditions which may confound quantifying postoperative pain resulting from surgery
* Current chronic opioid or tramadol use
* History of alcohol or opioid abuse
* Known allergy to the study medications
* Pregnancy
* Any health condition requiring greater than 100 micrograms of fentanyl during anesthesia induction
* Treated with any acetaminophen-containing medication in the previous 8 hours
* Treated with MAO inhibitors within 10 days prior to surgery
* Inability to communicate with the investigators and hospital staff
* Known or impaired liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the difference in proportions of patients from each treatment group who avoid using any opioids following anesthesia emergence until recovery room discharge. | Day of Surgery

SECONDARY OUTCOMES:
A secondary endpoint for this investigation will be the total dose of fentanyl administered to the patient. | Day of Surgery
A secondary outcome for this investigation will be the total dose of morphine administered to the patient. | Day of Surgery
A secondary outcome for this investigation will be the total dose of ibuprophen administered to the patient. | Day of Surgery
A secondary outcome measure for this investigation will be the total dose of oxycodone administered to the patient. | Day of Surgery
A secondary outcome measure will be any surgeon-administered local anesthetics used for wound infiltration. | Day of Surgery
A secondary outcome measure for this study will be any recovery-room anti-emetics administered to the patient. | Day of Surgery
Patients will be asked at time of PACU discharge, "Overall, how would you rate the study treatments?" Responses will be on 0 to 3 scale where 0=poor and 3=excellent. | Day of Surgery
Patients will be asked at time of PACU discharge, "Overall, how would you rate the level of pain relief from study medication?" Responses will be on 0 to 3 scale where 0=poor and 3=excellent. | Day of Surgery
Adverse events | Up to one year postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center (Hillcrest and Thornton), San Diego, California, United States